CLINICAL TRIAL: NCT01344304
Title: Multicenter Randomized Controlled Trial of Combination Antiemetic Therapy With Aprepitant / Fosaprepitant in Patients With Colorectal Cancer Receiving Oxaliplatin-based Chemotherapy
Brief Title: Study of Aprepitant / Fosaprepitant for the Prevention of Chemotherapy-induced Nausea and Vomiting (CINV) in Colorectal Cancer Patients - SENRI Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Multicenter Clinical Study Group of Osaka, Colorectal Cancer Treatment Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SENRI
Record Dates: First submitted 2011-04-27; First posted 2011-04-29 (Estimated); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Colorectal Cancer
Keywords: aprepitant therapy; fosaprepitant therapy; 5HT3-receptor antagonist; dexamethasone; colorectal cancer; FOLFOX; XELOX; SOX
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Aprepitant; fosaprepitant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard therapy (No Intervention): The patients are treated with 5HT3-receptor antagonist + dexamethasone during the first course, then treated with aprepitant / fosaprepitant + 5HT3-receptor antagonist + dexamethasone
- Aprepitant / Fosaprepitant therapy (Experimental): The patients are treated with aprepitant / fosaprepitant + 5HT3-receptor antagonist + dexamethasone during first and second courses.
  Interventions: Drug: Aprepitant / Fosaprepitant

INTERVENTIONS:
Drug: Aprepitant / Fosaprepitant — Aprepitant:
  125 mg PO on day 1 80 mg PO on days 2 to 3
  Fosaprepitant:
  150 mg IV on day 1
  Arms: Aprepitant / Fosaprepitant therapy

SUMMARY:
The object of this study is to evaluate the superiority of aprepitant therapy with a 5HT3-receptor antagonist, dexamethasone and aprepitant compared to standard therapy with a 5HT3-receptor antagonist and dexamethasone for prevention of nausea and vomiting in first course chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥20 years old
* Sex: Not specified
* Patients with colon/rectal cancer who first underwent FOLFOX, XELOX or SOX regimen including oxaliplatin at ≥85 mg/m2 (naive patient), or those who had already started chemotherapy and had nausea of Grade 2 or higher in the last course or an earlier course (non-naive patient).
* Stage: not specified (neoadjuvant/adjuvant chemotherapy, advanced or recurrent type are allowed)
* Combination of molecular targeted therapy: allowable
* Written informed consent for participation in the study.

Exclusion Criteria:

* Severe liver or kidney disease
* Nausea/vomiting within 24 hr prior to chemotherapy.
* Treatment with antiemetics within 24 hr prior to chemotherapy.
* Presence of factors causing nausea/vomiting other than chemotherapy (e.g. brain tumor, gastrointestinal obstruction, active peptic ulcer disease, brain metastasis)
* Presence of a disease precluding 3-day administration of dexamethasone (e.g. uncontrollable diabetes)
* Pregnant or lactating women, women who plan to become pregnant.
* Current treatment with pimozide.
* Any patient judged to be inappropriate for the study by the investigator.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 413 (Actual)
Dates: Start 2011-04; Primary Completion 2013-11 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Patient diary recording nausea, emesis, food ingestion, and rescue therapy | From initiating administration of anticancer agents to day 6 (120 hours)

CONTACTS AND LOCATIONS:
Locations (27):
- Japan (27):
  - Kansai Rosai Hospital, Amagasaki, Hyōgo
  - Kinki Central Hospital, Itami, Hyōgo
  - Kawasaki Hospital, Kobe, Hyōgo
  - Nara Hospital Kinki University Faculty of Medicine, Ikoma, Nara
  - Higashiosaka City General Hospital, Higashiosaka, Osaka
  - Saito Yukoukai Hospital, Ibaraki, Osaka
  - Rinku General Medical Center, Izumisano, Osaka
  - Kaizuka City Hospital, Kaizuka, Osaka
  - Hannan Chuo Hospital, Matsubara, Osaka
  - Minoh City Hospital, Minoo, Osaka
  - Sakai City Hospital, Sakai, Osaka
  - Osaka Rosai Hospital, Sakai, Osaka
  - Suita Municipal Hospital, Suita, Osaka
  - Saiseikai Senri Hospital, Suita, Osaka
  - Graduate School of Medicine / Faculty of Medicine, Osaka University, Suita, Osaka
  - Toyonaka Municipal Hospital, Toyonaka, Osaka
  - Yao Municipal Hospital, Yao, Osaka
  - Kenporen Osaka Central Hospital, Osaka
  - Iseikai Hospital, Osaka
  - Osaka Medical Center for Cancer and Cardiovascular Diseases, Osaka
  - National Hospital Organization Osaka National Hospital, Osaka
  - NTT West Osaka Hospital, Osaka
  - Nissay Hospital, Osaka
  - Tane General Hospital, Osaka
  - Osaka Seninhoken Hospital, Osaka
  - Osaka Koseinenkin Hospital, Osaka
  - Osaka General Medical Center, Osaka